CLINICAL TRIAL: NCT02105194
Title: Hyperbaric Oxygen Therapy and SPECT Brain Imaging in Cerebral Decompression Illness
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul G. Harch, M.D. (Other)
Collaborators: Harch Hyperbaric Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Paul G. Harch, M.D., Clinical Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Organization: Louisiana State University Health Sciences Center in New Orleans (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSU IRB #6627
Record Dates: First submitted 2014-03-30; First posted 2014-04-07 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Cerebral Decompression Illness, All Phases
Keywords: cerebral decompression illness
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric oxygen therapy (Experimental): Hyperbaric oxygen therapy
  Interventions: Drug: Hyperbaric oxygen therapy

INTERVENTIONS:
Drug: Hyperbaric oxygen therapy — total body exposure to greater than atmospheric pressure oxygen

SUMMARY:
Chart review of patients who received hyperbaric oxygen therapy for cerebral decompression illness who also underwent SPECT brain blood flow imaging to see if SPECT brain imaging tracks and is consistent with the clinical condition of the patients.

DETAILED DESCRIPTION:
SPECT brain imaging has been shown to be the most sensitive imaging modality for cerebral decompression illness. This study is a retrospective review of the PI's experience using SPECT brain imaging in the diagnosis and treatment of all phases of cerebral decompression illness over the past two decades. The purpose of the study is to see if the functional imaging is consistent with the clinical condition and cognitive testing. Chart review of symptoms, and physical exam findings will be compared before and after treatment to SPECT brain imaging radiological readings to assess concordance.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the P.I.'s practice who underwent hyperbaric oxygen therapy for cerebral decompression illness in the previous two decades who also underwent SPECT brain blood flow imaging early in the course of treatment and following completion of hyperbaric oxygen therapy.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
SPECT brain imaging | Within one month after completion of hyperbaric oxygen therapy
  Comparison of SPECT brain imaging chart copy of radiological reading before or early in the treatment history to SPECT brain imaging chart copy of radiological reading after treatment. Imaging will be scored as better, worse, or no change based on resolution of defects or improvement in pattern of injury.

SECONDARY OUTCOMES:
Symptoms of cerebral decompression illness | Within one month after hyperbaric oxygen therapy
  Chart reports of patients' symptoms of cerebral decompression illness before hyperbaric oxygen therapy will be compared to symptoms after hyperbaric oxygen therapy and rated as better, worse, or no change.
Abnormal physical exam findings | Within one month after hyperbaric oxygen therapy
  Chart reports of abnormal physical exam findings before hyperbaric oxygen therapy will be compared to chart reports of physical exam findings after hyperbaric oxygen therapy and rated as better, worse, or no change.

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Harch, M.D., Principal Investigator — LSU School of Medicine
Locations (1):
- Family Physicians Center, Marrero, Louisiana, United States